CLINICAL TRIAL: NCT05810636
Title: Hyperactivity Assessment in Children With Attention-deficit Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202110059RINB
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD group: Inclusion criteria:
  * DSM-5 Attention-deficit hyperactivity disorder
  * 7~18 years old
  * Willing to carry smartwatch and smartphone most of the time during one-month study period
  Exclusion criteria:
  - Comorbid with major psychiatric disorders (i.e., schizophrenia, bipolar disorder) or neurodevelopmental disorders (i.e., intellectual disability, autism spectrum disorder)
  Interventions: Device: Garmin Vivosmart wearable device
- Neurotypical group: Inclusion criteria:
  * 7~18 years old without a diagnosis of Attention-deficit hyperactivity disorder
  * Willing to carry smartwatch and smartphone most of the time during one-month study period
  Exclusion criteria:
  * Have a diagnosis of major psychiatric disorders (i.e., schizophrenia, bipolar disorder) or neurodevelopmental disorders (i.e., intellectual disability, autism spectrum disorder)
  * Unable to use smartwatch and smartphone
  Interventions: Device: Garmin Vivosmart wearable device

INTERVENTIONS:
Device: Garmin Vivosmart wearable device — Wearing smartwatches to collect data

SUMMARY:
Attention-deficit hyperactivity disorder (ADHD) is a neurodevelopmental disorder characterized by inattention, hyperactivity, and impulsivity. Clinical diagnosis of this disorder depends of history taking, parent report, and questionnaire. Attention test such as continuous performance test can provide quantitative measurement on attention deficits; however, there is a lack of objective tool to quantify the activity level. This study aims to assess activity level in children with ADHD. We plan to recruit 50 children with ADHD and 50 neurotypical children. The activity level measured by wearable device will be compared between ADHD and neurotypical children. The correlation between behavior rating on questionnaire and quantitative data measured by wearable device will be analyzed.

ELIGIBILITY:
ADHD group:

Inclusion criteria:

* DSM-5 Attention-deficit hyperactivity disorder
* 7~18 years old
* Willing to carry smartwatch and smartphone most of the time during one-month study period

Exclusion criteria:

* Comorbid with major psychiatric disorders (i.e., schizophrenia, bipolar disorder) or neurodevelopmental disorders (i.e., intellectual disability, autism spectrum disorder)
* Unable to use smartwatch and smartphone

Neurotypical group:

Inclusion criteria:

* 7~18 years old without a diagnosis of Attention-deficit hyperactivity disorder
* Willing to carry smartwatch and smartphone most of the time during one-month study period

Exclusion criteria:

* Have a diagnosis of major psychiatric disorders (i.e., schizophrenia, bipolar disorder) or neurodevelopmental disorders (i.e., intellectual disability, autism spectrum disorder)
* Unable to use smartwatch and smartphone

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Students from 1st grade to 12th grade who are eligible based on the criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceleration | 24 hours for 30 days
  Arm Acceleration

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton C, McKinstry B, Szentagotai Tatar A, Serrano-Blanco A, Pagliari C, Wolters M. Activity monitoring in patients with depression: a systematic review. J Affect Disord. 2013 Feb 15;145(1):21-8. doi: 10.1016/j.jad.2012.07.001. Epub 2012 Aug 4. PMID 22868056
- [Background] Cho CH, Lee T, Kim MG, In HP, Kim L, Lee HJ. Mood Prediction of Patients With Mood Disorders by Machine Learning Using Passive Digital Phenotypes Based on the Circadian Rhythm: Prospective Observational Cohort Study. J Med Internet Res. 2019 Apr 17;21(4):e11029. doi: 10.2196/11029. PMID 30994461
- [Background] Couronne R, Probst P, Boulesteix AL. Random forest versus logistic regression: a large-scale benchmark experiment. BMC Bioinformatics. 2018 Jul 17;19(1):270. doi: 10.1186/s12859-018-2264-5. PMID 30016950
- [Background] Dogan E, Sander C, Wagner X, Hegerl U, Kohls E. Smartphone-Based Monitoring of Objective and Subjective Data in Affective Disorders: Where Are We and Where Are We Going? Systematic Review. J Med Internet Res. 2017 Jul 24;19(7):e262. doi: 10.2196/jmir.7006. PMID 28739561
- [Background] Gau SS, Chen SJ, Chou WJ, Cheng H, Tang CS, Chang HL, Tzang RF, Wu YY, Huang YF, Chou MC, Liang HY, Hsu YC, Lu HH, Huang YS. National survey of adherence, efficacy, and side effects of methylphenidate in children with attention-deficit/hyperactivity disorder in Taiwan. J Clin Psychiatry. 2008 Jan;69(1):131-40. doi: 10.4088/jcp.v69n0118. PMID 18312048
- [Background] Gau SS, Lin CH, Hu FC, Shang CY, Swanson JM, Liu YC, Liu SK. Psychometric properties of the Chinese version of the Swanson, Nolan, and Pelham, Version IV Scale-Teacher Form. J Pediatr Psychol. 2009 Sep;34(8):850-61. doi: 10.1093/jpepsy/jsn133. Epub 2008 Dec 12. PMID 19074488
- [Background] Gau SS, Shang CY, Liu SK, Lin CH, Swanson JM, Liu YC, Tu CL. Psychometric properties of the Chinese version of the Swanson, Nolan, and Pelham, version IV scale - parent form. Int J Methods Psychiatr Res. 2008;17(1):35-44. doi: 10.1002/mpr.237. PMID 18286459
- [Background] Leikauf JE, Correa C, Bueno AN, Sempere VP, Williams LM. StopWatch: Pilot study for an Apple Watch application for youth with ADHD. Digit Health. 2021 Apr 1;7:20552076211001215. doi: 10.1177/20552076211001215. eCollection 2021 Jan-Dec. PMID 33868703
- [Background] Martin JL, Hakim AD. Wrist actigraphy. Chest. 2011 Jun;139(6):1514-1527. doi: 10.1378/chest.10-1872. PMID 21652563
- [Background] Marzano L, Bardill A, Fields B, Herd K, Veale D, Grey N, Moran P. The application of mHealth to mental health: opportunities and challenges. Lancet Psychiatry. 2015 Oct;2(10):942-8. doi: 10.1016/S2215-0366(15)00268-0. Epub 2015 Sep 29. PMID 26462228
- [Background] Patel MS, Foschini L, Kurtzman GW, Zhu J, Wang W, Rareshide CAL, Zbikowski SM. Using Wearable Devices and Smartphones to Track Physical Activity: Initial Activation, Sustained Use, and Step Counts Across Sociodemographic Characteristics in a National Sample. Ann Intern Med. 2017 Nov 21;167(10):755-757. doi: 10.7326/M17-1495. Epub 2017 Sep 26. No abstract available. PMID 28973116
- [Background] Polanczyk G, de Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry. 2007 Jun;164(6):942-8. doi: 10.1176/ajp.2007.164.6.942. PMID 17541055
- [Background] Reinertsen E, Clifford GD. A review of physiological and behavioral monitoring with digital sensors for neuropsychiatric illnesses. Physiol Meas. 2018 May 15;39(5):05TR01. doi: 10.1088/1361-6579/aabf64. PMID 29671754
- [Background] Simon V, Czobor P, Balint S, Meszaros A, Bitter I. Prevalence and correlates of adult attention-deficit hyperactivity disorder: meta-analysis. Br J Psychiatry. 2009 Mar;194(3):204-11. doi: 10.1192/bjp.bp.107.048827. PMID 19252145
- [Background] Swanson JM, Kraemer HC, Hinshaw SP, Arnold LE, Conners CK, Abikoff HB, Clevenger W, Davies M, Elliott GR, Greenhill LL, Hechtman L, Hoza B, Jensen PS, March JS, Newcorn JH, Owens EB, Pelham WE, Schiller E, Severe JB, Simpson S, Vitiello B, Wells K, Wigal T, Wu M. Clinical relevance of the primary findings of the MTA: success rates based on severity of ADHD and ODD symptoms at the end of treatment. J Am Acad Child Adolesc Psychiatry. 2001 Feb;40(2):168-79. doi: 10.1097/00004583-200102000-00011. PMID 11211365
- [Background] Tazawa Y, Wada M, Mitsukura Y, Takamiya A, Kitazawa M, Yoshimura M, Mimura M, Kishimoto T. Actigraphy for evaluation of mood disorders: A systematic review and meta-analysis. J Affect Disord. 2019 Jun 15;253:257-269. doi: 10.1016/j.jad.2019.04.087. Epub 2019 Apr 22. PMID 31060012